CLINICAL TRIAL: NCT00164801
Title: Is Visceral Hyperalgesia the Culprit of Noncardiac Chest Pain in Chinese? Part 2: Effect of GABAB Agonist on Visceral Hyperalgesia in NCCP Patients
Brief Title: Effect of GABAB Agonist on Visceral Hyperalgesia in NCCP patientsChinese?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPB study
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Non-Cardiac Chest Pain
MeSH Terms: interventions — Baclofen; Diltiazem

INTERVENTIONS:
Drug: Baclofen, Diltiazem

SUMMARY:
The effect of baclofen (GABAB agonist), diltiazem (muscle relaxant) and placebo will be compared in a double-blinded randomized study for the treatment of NCCP. Cerebral cortical, brainstem and spinal evoked potentials before and after treatment will be evaluated. Results of this study will shed lights on pathogenesis and treatment of NCCP in Chinese.We hypothesize that Baclofen alleviates visceral hyperalgesia in NCCP patients by suppressing afferent sensory pathway.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with monthly angina-like chest pain and negative coronary angiogram or scintigraphy
* Age between 18-70
* Gastroesophageal reflux disease
* Psychiatric illness
* Cerebrovascular accident
* Active peptic ulceration
* Heart failure or cardiac bradyarrhythmia
* Epilepsy
* Pregnancy or lactating female
* Previous hypersensitivity to muscle relaxant

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-11; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Esophageal sensory and pain thresholds

SECONDARY OUTCOMES:
Symptom severity of chest pain at the end of treatment
Evoked potential responses

CONTACTS AND LOCATIONS:
Overall Officials: Justin CY CU, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, China